CLINICAL TRIAL: NCT04093362
Title: A Phase 3, Open-Label, Randomized Study of Futibatinib Versus Gemcitabine-Cisplatin Chemotherapy as First-Line Treatment of Patients With Advanced Cholangiocarcinoma Harboring FGFR2 Gene Rearrangements FOENIX-CCA3
Brief Title: Futibatinib Versus Gemcitabine-Cisplatin Chemotherapy as First-Line Treatment of Patients With Advanced Cholangiocarcinoma Harboring FGFR2 Gene Rearrangements
Acronym: FOENIX-CCA3
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to Poor Recruitment
Sponsor: Taiho Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAS-120-301; 2019-004630-42 (EudraCT Number)
Record Dates: First submitted 2019-09-16; First posted 2019-09-18 (Actual); Results first posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Advanced Cholangiocarcinoma; FGFR2 Gene Rearrangements
Keywords: Futibatinib; Advanced Cholangiocarcinoma; FGFR2; Fusion; Rearrangement; TAS-120
MeSH Terms: interventions — futibatinib; Cisplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Futibatinib (Experimental): Participants received futibatinib at an oral dose of 20 milligrams (mg), administered once daily (QD) on every day of a 21-day cycle up to disease progression.
  Interventions: Drug: Futibatinib
- Cisplatin/Gemcitabine (Active Comparator): Participants received cisplatin 25 milligrams per square meter (mg/m^2) IV infusion followed by gemcitabine 1000 mg/m^2 IV infusion on Days 1 and 8 of each 21-day cycle up to 8 cycles.
  Interventions: Drug: Cisplatin; Drug: Gemcitabine

INTERVENTIONS:
Drug: Futibatinib — Oral tablets
  Other Names: TAS-120
  Arms: Futibatinib
Drug: Cisplatin — IV infusion
  Arms: Cisplatin/Gemcitabine
Drug: Gemcitabine — IV infusion
  Arms: Cisplatin/Gemcitabine

SUMMARY:
This is an open-label, multinational, parallel 2-arm, randomized Phase 3 study evaluating the efficacy and safety of futibatinib versus gemcitabine-cisplatin chemotherapy as first-line treatment of participants with advanced, metastatic, or recurrent unresectable intrahepatic cholangiocarcinoma (iCCA) harboring FGFR2 gene rearrangements

DETAILED DESCRIPTION:
Study TAS-120-301 is an open-label, multinational, parallel 2-arm, randomized Phase 3 study evaluating the efficacy and safety of futibatinib versus gemcitabine-cisplatin chemotherapy as first-line treatment of participants with advanced, metastatic, or recurrent unresectable iCCA harboring FGFR2 gene rearrangements. Eligible participants will be randomized on a 1:1 basis to the following study arms:

* Experimental Arm: Participants will receive futibatinib at an oral dose of 20 mg, administered daily (QD) on every day of a 21-day cycle.
* Control Arm: On Days 1 and 8 of a 21-day cycle, participants will receive:

  * Cisplatin 25 mg/m2 in 1000 mL 0.9% saline by intravenous (IV) infusion over 1 hour, followed by 500 millilliteres (mL) 0.9 percent (%) saline over 30 minutes; and
  * Gemcitabine 1000 mg/m2 in 250-500 mL 0.9% saline by IV infusion over 30 minutes, beginning after completion of the cisplatin and saline infusions.

Participants in the Experimental Arm may continue to receive continuous futibatinib until documentation of progressive disease (PD) per Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v 1.1), or until other withdrawal criteria are met, whichever comes first. However, treatment may continue following PD per RECIST 1.1 if the participants is clinically stable and is considered by the Investigator to be deriving continued clinical benefit from futibatinib.

Participants in the Control Arm may receive gemcitabine-cisplatin chemotherapy for up to 8 cycles or until PD or other withdrawal criteria are met, whichever comes first. Participants who discontinue gemcitabine-cisplatin due to documented disease progression (by ICR) may receive treatment with futibatinib ("crossover"), if medically appropriate in the opinion of the Investigator and if criteria for futibatinib treatment are met.

ELIGIBILITY:
Inclusion Criteria:

A participant must meet all of the following inclusion criteria to be eligible for enrollment in this study:

1. Provide written informed consent.
2. Is ≥18 years of age (or meets the country's regulatory definition for legal adult age).
3. The participant has histologically confirmed, locally advanced, or metastatic, or recurrent unresectable iCCA harboring FGFR2 gene rearrangements based on testing performed by the designated central laboratory.
4. Participant has radiographically measurable disease per RECIST 1.1.
5. Participants who have received treatment for locally advanced disease (for example, trans-arterial chemoembolization, selective internal radiation therapy, external beam radiation) must have evidence of radiographic progression with measurable disease outside the previously-treated lesions.
6. Eastern Cooperative Oncology Group performance status (ECOG PS) 0 or 1.
7. Adequate organ function as defined by the following criteria:

   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3.0 ×upper limit of normal (ULN); if liver function abnormalities are due to underlying liver metastasis, AST and ALT ≤ 5 × ULN.
   * Total bilirubin ≤ 1.5 × ULN, or ≤ 3.0 × ULN for participants with Gilbert's syndrome.
   * White Blood Count (WBC) ≥ 2000/mm3 (≥ 2.0 × 109/L)
   * Absolute neutrophil count (ANC) ≥ 1000/mm3 (ie, ≥ 1.0 × 109/L by International Units [IU])
   * Platelet count ≥ 100,000/mm3 (IU: ≥ 100 × 109/L)
   * Hemoglobin ≥ 9.0 g/dL
   * Phosphorus ≤ 1.5 × ULN
   * Creatinine clearance: ≥ 60 mL/min
8. Women of child-bearing potential (WOCBP) must have a negative serum pregnancy test within 7 days prior to administration of the first dose of futibatinib. Female participants are not considered to be of child bearing potential if they have a history of hysterectomy or are post menopausal defined as no menses for 12 months without an alternative medical cause. Both males and females of reproductive potential must agree to use effective birth control during the study prior to the first dose and for 6 months after the last dose.
9. Willing and able to comply with scheduled visits and study procedures.

Exclusion Criteria:

A participant will be excluded from this study if any of the following criteria are met:

1. Participant has received previous systemic anticancer therapy.

   •Participants receiving adjuvant or neoadjuvant treatment and completed ≥6 months prior to randomization are eligible.
2. Participant has mixed hepatocellular carcinoma - iCCA disease.
3. History and/or current evidence of any of the following disorders:

   * Non-tumor related alteration of calcium-phosphorus homeostasis that is clinically significant in the opinion of the Investigator.
   * Ectopic mineralization/calcification, including but not limited to soft tissue, kidneys, intestine, or myocardia and lung, considered clinically significant in the opinion of the Investigator.
   * Retinal disorder confirmed by retinal examination and considered clinically significant in the opinion of the ophthalmologist.
4. History or current evidence of uncontrolled ventricular arrhythmias
5. Fridericia's corrected QT interval (QTcF) > 470 milliseconds (ms) on electrocardiogram (ECG) conducted during Screening.
6. Treatment with any of the following within the specified time frame prior to the first dose of study therapy, or failure to recover from side effects of these prior therapies:

   * Major surgery within the previous 4 weeks (the surgical incision should be fully healed prior to the first dose of study therapy).
   * Radiotherapy (any dose) for extended field within 4 weeks or limited field radiotherapy within 2 weeks, and/or has not recovered from acute impact of radiotherapy.
   * Participants with locoregional therapy, e.g. transarterial chemoembolization (TACE), selective internal radiotherapy (SIRT) or ablation within 4 weeks.
   * Any history of liver transplant.
7. A serious illness or medical condition(s) including, but not limited to, the following:

   * Brain metastases that are untreated or clinically or radiologically unstable (that is, have been stable for <1 month).
   * Known acute systemic infection.
   * Myocardial infarction, severe/unstable angina, or symptomatic congestive heart failure within the previous 6 months.
   * Chronic nausea, vomiting, or diarrhea considered to be clinically significant in the opinion of the Investigator.
   * Congenital long QT syndrome, or any known history of torsade de pointes, or family history of unexplained sudden death.
   * Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that in the judgment of the Investigator would make the participant inappropriate for entry into this study.
8. Participants with a history of another primary malignancy that is currently clinically significant, and has potential for metastases or currently requires active intervention.
9. Pregnant or breast-feeding female.
10. The participant is unable to take oral medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-01-06 (Actual); Primary Completion 2024-04-22 (Actual); Study Completion 2024-04-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (103):
- United States (8):
  - City of Hope National Medical Center, Duarte, California
  - Norton Cancer Institute Audubon Hospital Campus Medical Plaza, Louisville, Kentucky
  - New Mexico Cancer Care Alliance, Albuquerque, New Mexico
  - Utah Cancer Specialists, Salt Lake City, Utah
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Medical Oncology Associates, PS - Summit Cancer Centers, Spokane, Washington
  - Carbone Comprehensive Cancer Center, Madison, Wisconsin
  - Medical College of Wisconsin - Froedtert Hospital, Milwaukee, Wisconsin
- Argentina (2):
  - Fundacion Favaloro para la Docencia e Investigacion Medica, Buenos Aires, Buenos Aires F.D.
  - Hospital de Gastroenterologia Dr. C. Bonorino Udaondo, Buenos Aires, Buenos Aires F.D.
- Australia (3):
  - Newcastle Private Hospital, Newcastle, New South Wales
  - Flinders Medical Centre, Bedford Park, South Australia
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
- Belgium (4):
  - UZ Antwerpen, Edegem, Antwerpen
  - Algemeen Ziekenhuis AZ Sint-Maarten, Mechelen, Antwerpen
  - AZ Delta Roeselare, Roeselare, Flanders
  - CHC MontLégia, Liège, Liege
- Brazil (9):
  - IOP - Instituto de Oncologia do Parana, Curitiba, Paraná
  - Instituto Nacional de Cancer Jose Alencar Gomes da Silva - INCA, Rio de Janeiro, Rio de Janeiro
  - Instituto Americas, Rio de Janeiro, Rio de Janeiro
  - Cepho-Fm Abc, Santo André, São Paulo
  - Hospital de Base de Sao Jose do Rio Preto, São José do Rio Preto, São Paulo
  - Instituto do Cancer do Estado de Sao Paulo, São Paulo, São Paulo
  - Fundacao Antonio Prudente - A.C.Camargo Cancer Center, São Paulo, São Paulo
  - Hospital Municipal Vila Santa Catarina, São Paulo, São Paulo
  - Hospital Santa Marcelina HSM, São Paulo, São Paulo
- France (8):
  - Hopitaux Universitaires Paris Nord Val de Seine - Hopital Beaujon, Clichy
  - Centre Georges-Francois Leclerc, Dijon
  - Centre Hospitalier Universitaire de Grenoble, La Tronche
  - Centre Leon Berard, Lyon
  - CHRU Besancon, Montbéliard
  - CHU Reims, Reims
  - Institut de Cancerologie Strasbourg Europe ICAENS, Strasbourg
  - CHU de TOURS - Hopital Trousseau, Tours
- Germany (3):
  - Charite - Universitaetsmedizin Berlin, Berlin
  - Universitaetsmedizin Mainz, Mainz
  - Technische Universitaet Muenchen - Klinikum rechts der Isar, München
- Hong Kong (2):
  - The University of Hong Kong, Queen Mary Hospital, Hong Kong
  - The Chinese University of Hong Kong Prince of Wales Hospital, Shatin
- Italy (9):
  - Candiolo Cancer Institute - FPO IRCCS, Candiolo
  - Ospedale Versilia, Lucca
  - AOU di Cagliari, Monserrato
  - Ospedale Maggiore della Carita di Novara, Novara
  - Servizio Sanitario Regionale Emilia-Romagna - Azienda Ospedaliero-Universitaria di Parma Ospedale Maggiore, Parma
  - Policlinico Uni. Campus Bio-Medico, Roma
  - Azienda Ospedaliera Universitaria Senese Policlinico Le Scotte, Siena
  - AOUI Verona - Ospedale Borgo Roma, Verona
  - Azienda ULSS 8 Berica, Vicenza
- Japan (12):
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Chiba University Hospital, Chiba, Chiba
  - National Cancer Center Hospital East, Kashiwa-Shi, Chiba
  - National Hospital Organization Kyushu Cancer Center, Fukuoka, Fukuoka
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - Nagasaki University Hospital, Nagasaki, Nagasaki
  - Osaka city University Hospital, Osaka, Osaka
  - Osaka University Hospital, Suita-shi, Osaka
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - The Cancer Institute Hospital of JFCR, Koto-Ku, Tokyo
  - Kyorin University Hospital, Mitaka-shi, Tokyo
- Mexico (3):
  - Centro de Estudios y Prevencion del Cancer (CEPREC), Tuxtla Gutiérrez, Chiapas
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico City, MX
  - Hospital Universitario Jose Eleuterio Gonzalez, Monterrey, Nuevo León
- Radboud University Medical Center, Nijmegen, GA, Netherlands
- Peru (4):
  - Instituto Nacional de Enfermedades Neoplasicas (INEN), Surquillo, Lima region
  - Hospital Daniel Alcides Carrion, Bellavista, Provincia Constitucional del Callao
  - Hospital Goyeneche, Arequipa
  - Hospital Nacional Arzobispo Loayza, Lima
- Poland (2):
  - Centrum Medyczne HCP Sp. z o.o., Poznan, Greater Poland Voivodeship
  - Szpital Kliniczny Przemienienia Pańskiego UM im. Karola Marcinkowskiego w Poznaniu, Poznan, Woj. Wielkopolskie
- Portugal (3):
  - Fundacao Champalimaud, Lisbon
  - CUF Porto Hospital, Porto
  - Instituto Portugues de Oncologia do Porto, Porto
- South Korea (8):
  - Chonnam National University Hwasun Hospital, Hwasun, Jeollanam-do
  - Seoul National University Hospital, Jungni I Gu, Seoul
  - Asan Medical Center, Seoul, Seoul
  - Dong-A University Hospital, Busan
  - Kyungpook National University Hospital, Daegu
  - CHA Bundang Medical Center, Seongnam
  - Yonsei University Health System - Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
- Spain (8):
  - Onkologikoa, Donostia / San Sebastian, Gipuzkoa
  - Hospital Universitario Virgen de la Arrixaca HUVA, El Palmar, Murcia
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Clinica Universidad de Navarra, Madrid
  - MD Anderson Cancer Center, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Clinica Universidad de Navarra, Pamplona
- Taiwan (6):
  - Chang Gung Memorial Hospital CGMH - Kaohsiung Branch, Kaohsiung City
  - Chang Gung Memorial Hospital, Linkou, Taichung
  - National Cheng Kung University Hospital NCKUH, Tainan
  - Chi Mei Medical Center CMMC - Yongkang branch, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- Thailand (5):
  - Songklanagarind Hospital, Faculty of Medicine, Prince of Songkla University, Hat Yai, Changwat Songkhla
  - Khon Kaen University KKU - Faculty of Medicine-Srinagarind Hospital, Khon Kaen, Muang
  - Chulabhorn Hospital, HRH Princess Chulabhorn College of Medical Science, Chulabhorn Royal Academy, Bangkok
  - Rajavithi hospital, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Faculty of Medicine, Chiang Mai University, Chiang Mai
- United Kingdom (3):
  - University Hospitals Bristol NHS Foundation Trust, Bristol
  - University College London Hospital NHS Foundation Trust, London
  - Royal Free London NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 10 participants took part in the study from 06 January 2021 to 22 April 2024.
Pre-assignment Details: Total 10 participants with advanced cholangiocarcinoma were enrolled & randomized to receive either futibatinib or gemcitabine-cisplatin. The study was later terminated by the sponsor due to poor recruitment.
Groups:
- Futibatinib: Participants received futibatinib at an oral dose of 20 milligrams (mg), administered once daily (QD) in each 21-day cycle up to a maximum of 649 days.
- Gemcitabine-Cisplatin: Participants received cisplatin 25 milligrams per square meter (mg/m^2) intravenous (IV) infusion followed by gemcitabine 1000 mg/m^2 IV infusion on Days 1 and 8 of each 21-day cycle up to a maximum of 155 days.
Period: Overall Study
Arm/Group | Futibatinib | Gemcitabine-Cisplatin
Started | 4 | 6
Completed | 0 | 0
Not Completed | 4 | 6
Not completed — Study Termination | 1 | 1
Not completed — Withdrawal of Consent | 1 | 0
Not completed — Death | 1 | 3
Not completed — Reason not Specified | 1 | 2

BASELINE CHARACTERISTICS:
Population: All Randomized Population included participants randomized to any treatment group in the study.
Groups:
- Futibatinib: Participants received futibatinib at an oral dose of 20 mg, administered QD in each 21-day cycle up to a maximum of 649 days.
- Gemcitabine-Cisplatin: Participants received cisplatin 25 mg/m^2 IV infusion followed by gemcitabine 1000 mg/m^2 IV infusion on Days 1 and 8 of each 21-day cycle up to a maximum of 155 days.
- Total: Total of all reporting groups
Arm/Group | Futibatinib | Gemcitabine-Cisplatin | Total
Number analyzed (Participants) | 4 | 6 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.3 (9.46) | 56.3 (12.77) | 61.5 (12.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5
  Male | 3 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 3 | 2 | 5
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 5 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time from date of randomization to the date of documentation of disease progression by independent central review (ICR), or date of death, whichever occurs first. Response assessments were made based on Response Evaluation Criteria in Solid Tumors (RECIST) guidelines (version 1.1, 2009)
Time Frame: Up to approximately 28 months
Population: As pre-specified in protocol, a total of 162 PFS events were required to perform PFS analysis. As only 10 participants were enrolled in this study, hence no data was collected or analyzed as planned for this outcome measure.
Arm/Group | Futibatinib | Gemcitabine-Cisplatin
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the proportion of participants experiencing a best overall response of partial response (PR) or complete response (CR) as per RECIST 1.1, based on ICR. PR was defined as at least a 30% decrease in the sum of diameters of the target lesions, taking as a reference the baseline sum diameters and persistence of one or more non-target lesion(s) and/or maintenance of tumor marker level above the normal limits. CR was defined as disappearance of all target lesions. Any pathological lymph node must have reduction in short axis to less than (<)10 millimeters (mm) and disappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (<10-mm short axis)
Time Frame: Up to approximately 28 months
Population: The data for this outcome measure was not collected or analyzed as planned because the study was terminated early due to poor recruitment.
Arm/Group | Futibatinib | Gemcitabine-Cisplatin
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR was defined as the proportion of participants experiencing a best overall response of stable disease (SD), PR or CR as per RECIST 1.1, based on central assessment of radiologic images. PR was defined as at least a 30% decrease in the sum of diameters of the target lesions, taking as a reference the baseline sum diameters and persistence of one or more non-target lesion(s) and/or maintenance of tumor marker level above the normal limits. CR was defined as disappearance of all target lesions. Any pathological lymph node must have reduction in short axis to <10 mm and disappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (<10-mm short axis).
Time Frame: Up to approximately 28 months
Population: as for outcome 2
Arm/Group | Futibatinib | Gemcitabine-Cisplatin
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of randomization until the date of death due to any cause.
Time Frame: Up to approximately 28 months
Population: as for outcome 2
Arm/Group | Futibatinib | Gemcitabine-Cisplatin
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Progression-Free Survival (PFS) Per Investigator Assessment
Description: PFS per investigator assessment is defined as the time from date of randomization to the date of disease progression based on investigator assessment of radiographic images or death, whichever occurs first.
Time Frame: Up to approximately 28 months
Population: As pre-specified in protocol, a total of 162 PFS events were required to perform PFS analysis. As only 10 participants were enrolled in this study, hence no data was collected for this outcome measure.
Arm/Group | Futibatinib | Gemcitabine-Cisplatin
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs), and Serious Adverse Events (SAEs)
Description: An adverse event (AE) was defined as any untoward medical condition in clinical investigation participant administered drug; it does not necessarily have to have causal relationship with this treatment. A TEAE was defined as an AE that started or worsened at the time of or after first dose of study drug administration and within 30 days after last dose of study drug and does not necessarily have a causal relationship to use of the study drug. TEAEs were assessed by Common Terminology Criteria for Adverse Events Version 5.0 (CTCAE v5.0). SAE was any untoward medical occurrence that at any dose: results in death, is life-threatening, required in participant hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is congenital anomaly/birth defect, important medical event. TEAEs included any clinically significant changes in clinical laboratory tests, vital signs, ophthalmological exams, and 12-lead electrocardiogram (ECG).
Time Frame: Up to approximately 28 months
Population: All Treated Population included all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Futibatinib | Gemcitabine-Cisplatin
Number analyzed (Participants) | 4 | 5
Participants
  TEAEs | 4 | 5
  SAEs | 2 | 3

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to end of study (Up to approximately 28 months)
Description: All Treated Population included all participants who received at least one dose of study drug.
Arm/Group | Futibatinib | Gemcitabine-Cisplatin
All-Cause Mortality (participants affected / at risk) | 1/4 | 3/5
Serious Adverse Events (participants affected / at risk) | 2/4 | 3/5
Other Adverse Events (participants affected / at risk) | 4/4 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Futibatinib (N=4) | Gemcitabine-Cisplatin (N=5)
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Abdominal sepsis (Infections and infestations) | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
General physical health deterioration (General disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Futibatinib (N=4) | Gemcitabine-Cisplatin (N=5)
Diarrhoea (Gastrointestinal disorders) | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 3
Ascites (Gastrointestinal disorders) | 1 | 2
Stomatitis (Gastrointestinal disorders) | 1 | 0
COVID-19 (Infections and infestations) | 1 | 0
Paronychia (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 1
Blood follicle stimulating hormone decreased (Investigations) | 1 | 0
Lipase increased (Investigations) | 1 | 1
Neutrophil count decreased (Investigations) | 1 | 1
Platelet count decreased (Investigations) | 1 | 1
Weight decreased (Investigations) | 1 | 0
Weight increased (Investigations) | 1 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 3 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 2
Hypochloraemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0
Onycholysis (Skin and subcutaneous tissue disorders) | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Ocular hyperaemia (Eye disorders) | 1 | 0
Serous retinopathy (Eye disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 5
Constipation (Gastrointestinal disorders) | 0 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Asthenia (General disorders) | 1 | 1
Face oedema (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 2
Influenza like illness (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 0 | 3
Mucosal inflammation (General disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 3
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Atrioventricular block second degree (Cardiac disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 2
International normalised ratio increased (Investigations) | 0 | 1
White blood cell count decreased (Investigations) | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 2
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1
Retinal haemorrhage (Eye disorders) | 0 | 1
Visual impairment (Eye disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Phlebitis (Vascular disorders) | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
The data for the outcome measures related to PFS, OS, ORR, DCR, and PFS per Investigator assessment was not collected or analyzed as planned because the study was terminated early due to poor recruitment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-01-29): https://cdn.clinicaltrials.gov/large-docs/62/NCT04093362/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-26): https://cdn.clinicaltrials.gov/large-docs/62/NCT04093362/SAP_001.pdf